CLINICAL TRIAL: NCT03076268
Title: Treinta Millones de Palabras-Visitas al Hogar Pilot Randomized Controlled Trial
Brief Title: TMP-Visitas al Hogar
Acronym: TMP-HV RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16-1579
Record Dates: First submitted 2017-03-02; First posted 2017-03-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Language Development

STUDY DESIGN:
Intervention Model Description: The investigators will deliver the TMP Curriculum to 45 Treatment families. The TMP Curriculum is comprised of 1) 12 educational modules, 2) animations and videos of real parent-child interactions to teach parents about the science behind child brain development, and model strategies for improving parents' child-directed speech, 3) video modeling and collaborative goal setting, and 4) quantitative linguistic feedback from Language ENvironment Analysis (LENA) recordings.
Who Masked: Participant
Masking Description: Participants will not be aware of which condition they are enrolled in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): The investigators will deliver the TMP Curriculum to 45 Treatment families. The TMP Curriculum is comprised of 1) 12 educational modules, 2) animations and videos of real parent-child interactions to teach parents about the science behind child brain development, and model strategies for improving parents' child-directed speech, 3) video modeling and collaborative goal setting, and 4) quantitative linguistic feedback from Language ENvironment Analysis (LENA) recordings. This curriculum is delivered in Spanish.
  Interventions: Behavioral: Treinta Millones de Palabras - Visitas al Hogar
- Control Group (No Intervention): The investigators will deliver a Nutrition Curriculum to 45Control families. The Nutrition Curriculum provides information about the importance of healthy nutrition for child development, strategies for healthy eating, and meal preparation.This curriculum is delivered in Spanish.

INTERVENTIONS:
Behavioral: Treinta Millones de Palabras - Visitas al Hogar — TMP-Visitas al Hogar is a cultural and linguistic adaptation of the TMW-Home Visiting curriculum into Spanish. The 12-module curriculum has been translated into Spanish and adapted to address concerns that are vital to mono- and bilingual Spanish-speaking families, including the broadening research base for when to introduce a second language to a child and the benefits of bilingualism.
  Arms: Treatment Group

SUMMARY:
Treinta Millones de Palabras- Visitas al Hogar (TMP) is designed to intervene upon mothers' knowledge, beliefs, and behavior, which in turn influences their interaction with their children, impacting children's development. The investigators will measure change in mothers' knowledge, beliefs, and behavior during and after intervention, and measure impacts on children's development across major developmental domains. Specifically, the investigators will measure mothers'

1. Knowledge of child language development and the role of parents in that development
2. Beliefs about the malleability of intelligence and their role in shaping their children's intelligence
3. Interaction with their child, specifically their linguistic input and responsiveness to their child's communication

Concurrently, the investigators will measure children's

1. Emergent oral language development, in both Spanish and English
2. Social-emotional development
3. Math and spatial reasoning skill development

ELIGIBILITY:
Inclusion Criteria:

* participants (i.e. parents and their children) who live at or below 200% of the federal poverty line,
* female caregivers with a child between the ages of 24-30 months old,
* participants whose preferred home language is Spanish,
* education level is less than or equal to a bachelor's degree.

Exclusion Criteria:

* participants (i.e. parents and their children) who live over 200% of the federal poverty line,
* parents under the age of 18,
* non-female primary care giver
* children younger than 24 months old or older than 30 months old (at start of study),
* parents who do not have legal custody of their child,
* parents whose child does not live with them,
* parents who are not with their child at least two full days per week,
* parents who are unable to commit to the intervention requirements,
* foster parents,
* children with significant cognitive or physical impairments, (specifically Autism Spectrum Disorder, Epilepsy, Cerebral Palsy, hearing impairment, Down Syndrome and blindness),
* parents who have earned or are currently working toward a graduate or professional degree (e.g. M.A., M.S., M.B.A), and
* parents whose preferred home language is not Spanish.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline LENA scores in Adult Word Count, Conversational Turn Count, and Child Vocalizations in month 12, data aggregated by treatment group. | Baseline, 12 months

SECONDARY OUTCOMES:
Change from baseline in parent knowledge about child development using the SPEAK survey in month 12, data aggregated by treatment group. | Baseline, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Thirty Million Words® Initiative at the University of Chicago Medicine, Chicago, Illinois, United States

REFERENCES:
- [Background] Suskind DL, Leffel KR, Graf E, Hernandez MW, Gunderson EA, Sapolich SG, Suskind E, Leininger L, Goldin-Meadow S, Levine SC. A parent-directed language intervention for children of low socioeconomic status: a randomized controlled pilot study. J Child Lang. 2016 Mar;43(2):366-406. doi: 10.1017/S0305000915000033. Epub 2015 Jun 4. PMID 26041013
- [Derived] List JA, Pernaudet J, Suskind DL. Shifting parental beliefs about child development to foster parental investments and improve school readiness outcomes. Nat Commun. 2021 Oct 1;12(1):5765. doi: 10.1038/s41467-021-25964-y. PMID 34599167
- See also: Click here for more information about the Thirty Million Words — https://tmwcenter.uchicago.edu/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT03076268/Prot_SAP_002.pdf